CLINICAL TRIAL: NCT02259894
Title: Safety, Pharmacokinetics, and Pharmacodynamics of Single Rising Oral Doses of BIRT 2584 XX (5, 30, 100, 200, 350, 500, and 700 mg) as a Solution in PEG 400 Administered to Healthy Male Volunteers. Placebo Controlled and Blinded at Each Dose Level.
Brief Title: Safety, Pharmacokinetics, and Pharmacodynamics of BIRT 2584 XX in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1206.1
Record Dates: First submitted 2014-10-07; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- BIRT 2584 (Experimental): single rising doses
  Interventions: Drug: BIRT 2584 XX
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIRT 2584 XX
  Arms: BIRT 2584
Drug: Placebo
  Arms: Placebo

SUMMARY:
To assess safety, tolerability, pharmacokinetics, and pharmacodynamics of BIRT 2584 XX in single rising oral doses of 5 mg to 700 mg in a polyethylene glycol 400 (PEG 400) solution in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >=18 and <=50 years
* BMI >=18.5 and <=29.9 kg/m2

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, haematological, oncological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Relevant history of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (< 1 month prior to administration or during the trial)
* Use of any drugs, which might influence the results of the trial, (< 10 days prior to study drug administration or expected during the trial)
* Participation in another trial with an investigational drug (< 2 months prior to administration or expected during trial)
* Smoker (> 10 cigarettes or >3 cigars or >3 pipes/day)
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation or loss > 400 mL, < 1 month prior to administration or expected during the trial
* Clinically relevant laboratory abnormalities
* Any ECG value outside of the reference range and of clinical relevance including, but not limited to QRS interval > 110 ms or QT interval, Bazett correction (QTcB) > 450 ms or QT interval >500 ms
* Inability to comply with dietary regimen of study centre
* Inability to comply with investigator's instructions

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2004-03; Primary Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 16 days after drug administration
Number of participants with clinically significant changes in vital signs | Up to 16 days after drug administration
Number of participants with abnormal changes in clinical laboratory parameters | Up to 16 days after drug administration
Number of participants with abnormal findings in 12-lead ECG (electrocardiogram) | Up to 16 days after drug administration
Number of participants with abnormal findings in physical examination | Screening and up to 16 days after drug administration

SECONDARY OUTCOMES:
Cmax (maximum concentration in plasma) | Up to 360 hours after drug administration
tmax (time from dosing to maximum concentration) | Up to 360 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time) interval from 0 extrapolated to infinity) | Up to 360 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time) interval from 0 to the last quantifiable analyte plasma concentration) | Up to 360 hours after drug administration
λz (terminal rate constant in plasma) | Up to 360 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | Up to 360 hours after drug administration
MRT(mean residence time of the analyte in the body) | Up to 360 hours after drug administration
CL/F (apparent oral clearance in plasma after oral administration) | Up to 360 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz) dose) | Up to 360 hours after drug administration
Ae0-48 (amount of analyte that is eliminated in urine from 0-48 hours) | Up to 48 hours after drug administration
fe0-48 (fraction of analyte eliminated in urine from 0-48 hours) | Up to 48 hours after drug administration
CLR,0-48 (renal clearance of the analyte from 0-48 hours) | Up to 48 hours after drug administration
Receptor occupancy as determined by binding of anti-LFA-1 antibody fragment (Fab) | Up to 360 hours after drug administration
Inhibition of IL-2 production | Up to 360 hours after drug administration
  in response to superantigen challenge ex vivo